CLINICAL TRIAL: NCT02814318
Title: Intrapartum Effect of Vancomycin on Rectovaginal GBS Colonization
Status: Terminated | Type: Observational
Why Stopped: Ancef (Cefazolin) became the new standard of care (instead of Vancomycin) for GBS prophylaxis if the patient is allergic to penicillin.
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 16-008
Record Dates: First submitted 2016-06-09; First posted 2016-06-27 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Group B Streptococcal Infection
Keywords: Vancomycin; Penicillin; Clindamycin; Group B streptococcal infection; Rectovaginal GBS colonization; Vaginal GBS colonization; Intrapartum; Prophylaxis
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IV Vancomycin: GBS positive laboring women who are allergic to penicillin and clindamycin and are treated using IV vancomycin.
  Interventions: Biological: Vaginal and rectovaginal swab cultures
- IV Penicillin: GBS positive laboring women who are not allergic to penicillin and are treated using IV penicillin.
  Interventions: Biological: Vaginal and rectovaginal swab cultures

INTERVENTIONS:
Biological: Vaginal and rectovaginal swab cultures — The only intervention that will occur in this study is obtaining vaginal and recto-vaginal swab cultures upon admission to the labor and delivery room and every two hours to follow until 8 hours after administration of IV vancomycin or IV penicillin.

SUMMARY:
The aim of this project is to identify the duration of vancomycin administration at which group B streptococcus (GBS) colonization is eradicated from the vaginal and recto-vaginal mucosa. This will aid in labor management and delivery planning to ensure that the mother receives adequate GBS prophylaxis while also minimizing the duration of exposure to vancomycin. In addition, this could prevent unnecessary prolonged hospitalization or septic workup of neonates whose mothers received vancomycin intrapartum.

This study aims to identify the time after administration of IV vancomycin at which GBS colonies are 100% eradicated.

DETAILED DESCRIPTION:
Prophylaxis of group B streptococcus has been a major component of prenatal care in preventing early onset of neonatal sepsis. While penicillin remains the gold standard medication for prophylaxis, this medication is not an option in women who have high risk allergic reactions to this class of medications. Furthermore, with rising rates of antibiotic resistance to erythromycin and clindamycin, more women are requiring vancomycin for GBS prophylaxis. While the CDC and ACOG recommend vancomycin as an alternative to penicillin for GBS prophylaxis, little research has been conducted investigating the transplacental passage of vancomycin.

Because of the gap in knowledge regarding intrapartum effects of IV vancomycin on GBS colonization, neonates of women who received vancomycin are considered as inadequately treated for GBS prophylaxis, and subsequently undergo additional observation, prolonged hospitalization, and possible septic workup in the immediate postpartum period. Because of this gap in knowledge, this research study investigates how quickly vaginal and recto-vaginal GBS colonization is eradicated to aid in timing of delivery in patients with GBS colonization who require vancomycin intrapartum.

In addition, the studies that investigated the duration of time of IV penicillin and IV clindamycin necessary for eradication of GBS colonization only investigated vaginal colonization, not recto-vaginal colonization. Their rationale was based on the assumption that most cases of neonatal GBS sepsis are caused by vaginal colonization. Given that the standard of care for GBS screening includes screening for colonization of both vaginal and rectal mucosa, investigators also plan to compare rates of eradication of GBS in vaginal colonies compared to recto-vaginal colonies.

ELIGIBILITY:
Vancomycin Arm

Inclusion Criteria

* Women aged 18 years or older
* Pregnancies of at least 37w0d gestation at delivery
* History of high-risk allergy to penicillin (including pruritic rash, urticaria, swelling, anaphylaxis)
* Women who are GBS positive
* Culture proven resistance or
* Unknown resistance to clindamycin or erythromycin

Exclusion Criteria

* Women with low risk allergy to penicillin
* History of allergy to vancomycin
* History of Red Man Syndrome
* History of renal or hepatic disease
* Immunocompromised patients
* History of chronic steroid use in current pregnancy
* Patient with fever or signs of chorioamnionitis on admission

Penicillin Arm

Inclusion Criteria

* Women aged 18 years or older
* Women who are GBS positive
* Pregnancies of at least 37w0d gestation at delivery

Exclusion Criteria

* Immunocompromised patients
* History of chronic steroid use in current pregnancy
* Patient with fever or signs of chorioamnionitis on admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: GBS positive laboring women aged at least 18 years old with pregnancies of 37 weeks gestational age or greater.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-06; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
GBS colonization levels after admission to labor and delivery | At 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: William Kim Brady, MD, Principal Investigator — TriHealth Inc.
Locations (2):
- United States (2):
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paccione KA, Wiesenfeld HC. Guideline adherence for intrapartum group B streptococci prophylaxis in penicillin-allergic patients. Infect Dis Obstet Gynecol. 2013;2013:917304. doi: 10.1155/2013/917304. Epub 2013 Feb 12. PMID 23476109
- [Background] Knight KM, Thornburg LL, McNanley AR, Hardy DJ, Vicino D, Glantz JC. The effect of intrapartum clindamycin on vaginal group B streptococcus colony counts. J Matern Fetal Neonatal Med. 2012 Jun;25(6):747-9. doi: 10.3109/14767058.2011.591458. Epub 2011 Jul 22. PMID 21780879
- [Background] McNanley AR, Glantz JC, Hardy DJ, Vicino D. The effect of intrapartum penicillin on vaginal group B streptococcus colony counts. Am J Obstet Gynecol. 2007 Dec;197(6):583.e1-4. doi: 10.1016/j.ajog.2007.08.045. PMID 18060942
- [Background] Turrentine MA, Greisinger AJ, Brown KS, Wehmanen OA, Mouzoon ME. Duration of intrapartum antibiotics for group B streptococcus on the diagnosis of clinical neonatal sepsis. Infect Dis Obstet Gynecol. 2013;2013:525878. doi: 10.1155/2013/525878. Epub 2013 Mar 28. PMID 23606801
- [Background] Laiprasert J, Klein K, Mueller BA, Pearlman MD. Transplacental passage of vancomycin in noninfected term pregnant women. Obstet Gynecol. 2007 May;109(5):1105-10. doi: 10.1097/01.AOG.0000260388.78339.b6. PMID 17470590
- [Background] Onwuchuruba CN, Towers CV, Howard BC, Hennessy MD, Wolfe L, Brown MS. Transplacental passage of vancomycin from mother to neonate. Am J Obstet Gynecol. 2014 Apr;210(4):352.e1-352.e4. doi: 10.1016/j.ajog.2014.01.019. PMID 24679944